CLINICAL TRIAL: NCT01900054
Title: A Long-Term Study of TAU-284 in Pediatric Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAU-284-18
Record Dates: First submitted 2013-07-03; First posted 2013-07-16 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Perennial Allergic Rhinitis
Keywords: TAU-284; Bepotastine besilate; Histamine H1 receptor antagonists; children
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — bepotastine besilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAU-284 (Experimental): Two TAU-284 5mg tablets will be taken orally twice a day, once after breakfast and once after dinner (or before bed).
  Interventions: Drug: Bepotastine besilate

INTERVENTIONS:
Drug: Bepotastine besilate — Two TAU-284 5mg tablets will be taken orally twice a day
  Other Names: TALION 5mg tablets

SUMMARY:
The objective of this study is to evaluate the long-term safety and efficacy of TAU-284 (Bepotastine besilate) in pediatric patients with perennial allergic rhinitis for 12 weeks administration.

DETAILED DESCRIPTION:
This is a multicenter,open-label, single-arm, uncontrolled study to evaluate the safety and efficacy of TAU-284 (20 mg/day) in pediatric patients with perennial allergic rhinitis for 12 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 and 15 years
* Patients who have received a diagnosis of perennial allergic rhinitis according to the diagnostic criteria
* Patients with a mean total score for the three major nasal symptoms [sneezing, rhinorrhea, and nasal congestion] of at least 3 on the basis of symptoms recorded in the nasal allergy diary during the observation period etc.

Exclusion Criteria:

* Patients with vasomotor rhinitis or eosinophilic rhinitis
* Patients who have concurrent nasal disease that may affect the efficacy of TAU-284
* Patients with a history of any of the nasal surgical procedures
* Patients with current or previous history of drug allergy
* Patients who concurrently have renal function abnormalities that may cause safety problems etc.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KIMIHIRO OKUBO, Study Director — Nippon Medical School
Locations (1):
- Reserch site, Kanagawa, Japan

REFERENCES:
- [Result] Okubo K, Ichimura M, Koyama T, Susuta Y, Izaki H. Double-blind placebo-controlled study of bepotastine besilate in pediatric patients with perennial allergic rhinitis. Expert Opin Pharmacother. 2015;16(16):2395-408. doi: 10.1517/14656566.2015.1085511. Epub 2015 Sep 12. PMID 26364765

RESULTS

PARTICIPANT FLOW:
Groups:
- TAU-284: TAU-284 10mg twice daily for 12 weeks
Period: Overall Study
Arm/Group | TAU-284
Started | 58
Completed | 56
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TAU-284
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events and Adverse Drug Reactions
Time Frame: Up to Week 12
Measure: Number; unit: participants
Arm/Group | TAU-284
Number analyzed (Participants) | 58
participants
  Adverse events | 37
  Adverse drug reactions | 2

2. Secondary Outcome: Change From Baseline in Total Score for the Three Major Nasal Symptoms [Sneezing, Rhinorrhea, and Nasal Congestion] at Week2, Week4, Week6, Week8, Week10, Week 12 and Final Evaluation Point.
Description: Total score for the three major nasal symptoms (sneezing, rhinorrhea, and nasal congestion) were rated on 5-point scale ranging from 0 (no symptom) to 4 (very severe).
Time Frame: Baseline, Week2, Week4, Week6, Week8, Week10, Week 12 and Final Evaluation Point （up to Week 12）
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | TAU-284
Number analyzed (Participants) | 58
units on a scale
  Week 2 | -0.943 (1.549)
  Week 4 | -1.388 (1.465)
  Week 6 | -1.321 (1.844)
  Week 8 | -1.433 (1.880)
  Week 10 | -1.460 (1.777)
  Week 12 | -1.451 (1.707)
  final evaluation point | -1.440 (1.678)

3. Secondary Outcome: Change From Baseline in Individual Nasal Symptom Scores (Sneezing, Rhinorrhea, Nasal Congestion, and Impairment in Daily Activities)
Time Frame: baseline, Week2, Week4, Week6, Week8, Week10 and Week 12
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Individual Scores for Local Nasal Findings (Rhinoscopic Findings)
Time Frame: Second enrollment, Week2, Week4, Week6, Week8, Week10 and Week 12
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Severity Score for Symptoms of Allergic Rhinitis
Time Frame: baseline, Week2, Week4, Week6, Week8, Week10 and Week 12
Reporting Status: Not Posted

6. Secondary Outcome: Influence of Activities in Daily Life(Study, Outing, Sleeping)
Time Frame: Second enrollment, Week2, Week4, Week6, Week8, Week10 and Week 12
Reporting Status: Not Posted

7. Secondary Outcome: Patient Impression of Nasal Symptoms(Sneezing, Rhinorrhea, Nasal Congestion, Nasal Pruritus, Eye Pruritus and Eye Tearing)
Time Frame: Week 12 or suspension
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | TAU-284
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 31/58
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAU-284 (N=58)
Nasopharyngitis (Infections and infestations) | 19
Otitis externa (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Liver function test abnormal (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other